CLINICAL TRIAL: NCT02684669
Title: Effect of High-dose Target-controlled Naloxone Infusion on Pain and Hyperalgesia During a Burn Injury. A Randomized, Placebo-controlled, Double-blind Crossover Study
Brief Title: Effect of High-dose Target-controlled Naloxone Infusion on Pain and Hyperalgesia During a Burn Injury
Acronym: TCI-NX-BI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: mads u werner (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, mads u werner, MD, DMSci, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-15018869-BI
Record Dates: First submitted 2016-02-10; First posted 2016-02-18 (Estimated); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Healthy Subjects
Keywords: burn injury; controlled trial; latent sensitization; naloxone; secondary hyperalgesia; volunteers
MeSH Terms: conditions — Burns; Hyperalgesia | interventions — Naloxone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-dose naloxone (Experimental): naloxone 4 mg/ml i.v. infusion, total 3.25 mg/kg, target controlled infusion with three infusion rates (0.25 mg/kg; 0.75 mg/kg; 2.25 mg/kg) each of 25 min duration.
  Interventions: Drug: Naloxone
- Normal saline (Placebo Comparator): 0.9% physiological saline, i.v. infusion, total 0.81 ml/kg, target controlled infusion with three infusion rates (0.06 ml/kg; 0.19 ml/kg; 0.56 ml/kg) each of 25 min duration.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Naloxone — active drug infusion
  Other Names: Naloxon "B. Braun"
  Arms: High-dose naloxone
Drug: Normal saline — placebo comparator
  Other Names: Physiologic Saline
  Arms: Normal saline

SUMMARY:
In several rodent studies, it has been demonstrated that very high doses of opioid antagonists (i.e., naloxone 3-10 mg/kg) administered after weeks after recovery from an inflammatory injury may lead to a reinstatement of hyperalgesia and pain behavior. This latent sensitization has recently been demonstrated also to take place in humans.

The present study examines if it is possible to foresee individuals who will demonstrate a larger degree of latent sensitization upon challenge with an injury, than others. Using an enriched design high sensitizers (e.g., the upper quartile of individuals developing large areas of secondary hyperalgesia following a mild burn injury) are compared with low sensitizers (lower quartile), regarding the propensity for developing latent sensitization

DETAILED DESCRIPTION:
Naloxone is a mu-opioid-receptor (MOR) antagonist drug, which dose-dependently exhibits hypo-algesic and hyper-algesic properties. Naloxone (and other MOR-antagonists) have been used in research to study the role of endogenous opioids in central processing of pain. It has been hypothesized that the endogenous opioid modulation of pain is impaired or altered in chronic pain conditions.

In a previous study using an electrical pain model in human patients, naloxone (21 microg/kg) increased the established area of secondary hyperalgesia. Further, administration of naloxone and naltrexone to animals following resolution of an inflammatory condition, have demonstrated a reinstatement of hypersensitivity to a noxious stimulus, indicating latent sensitization. It has thus been speculated that endogenous opioids may play an important role in the transition from acute to chronic pain in humans.

Recently, however, the investigators were unable to show reinstatement of secondary hyperalgesia after resolution of a burn injury by administrating naloxone in a low dose (21 microg/kg). Based on these finding the investigators hypothesized, that the negative results may be due to the low dose of naloxone or insufficient tissue injury to generate latent sensitization.

The systemic doses of opioid antagonists used in animal studies to demonstrate latent sensitization have been 0.3 to 3.0 mg/kg of naltrexone or 3-10 mg/kg of naloxone. Further, high doses of 1-2 mg/kg of naloxone have been used in clinical and experimental psychiatric, endocrinological, neurological and nutritional studies in patients and healthy individuals. In one pain related study, 6 mg/kg of naloxone was given to healthy patients intramuscularly. Only mild to moderate, transitory side-effects were recorded in these studies.

The investigators, therefore, initiated a second translational study in which it was hypothesized that a higher dose of naloxone (2 mg/kg) would reinstate secondary hyperalgesia in human patients following resolution of a mild burn injury and thus show latent sensitization in humans. The investigators demonstrated in 4 out of 12 patients that naloxone administered 7 days after a mild burn injury was associated with the reinstatement of secondary hyperalgesia.

The present study examines if it is possible to foresee individuals who will demonstrate a larger degree of latent sensitization upon challenge with an injury, than others. Using an enriched design high sensitizers (e.g., the upper quartile of individuals developing large areas of secondary hyperalgesia following a mild burn injury) are compared with low sensitizers (lower quartile), regarding the propensity for developing latent sensitization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Signed informed consent
* Urin-sample without traces of opioids (morphine, methadone, buprenorphine, codeine, tramadol, ketobemidone, oxycodone, hydromorphone, dextro-methorphan)
* ASA I
* Body mass index (BMI): 18 < BMI < 30 kg/sq.m

In addition Days 2-4:

• Secondary hyperalgesia areas 1 hr after a burn injury belonging to the upper quartile (Q3: high-sensitizers [n = 20]) or the lower quartile (Q1: low-sensitizers [n = 20]) The selection is made during a separate test day (Day 0 [n = 80]).

Exclusion Criteria:

* Participants, who do not speak or understand Danish
* Participants, who cannot cooperate with the investigation
* Allergic reaction against morphine or other opioids (including naloxone)
* Abuse of alcohol or drugs - according to investigator's evaluation
* Use of psychotropic drugs
* Neurologic or psychiatric disease
* Signs of neuropathy in the examination region
* Previous severe trauma to the lower legs with sequelae
* Scarring or tattoos in the examination areas
* Chronic pain condition
* Regular use of analgesic drugs
* Use of prescription drugs one week before the trial
* Use of over-the-counter (OTC) drugs 48 hours before the trial
* Does not develop measurable secondary hyperalgesia areas after BI

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Changes in areas of secondary hyperalgesia will be assessed before and after naloxone/placebo administration by a weighted-pin instrument | Baseline, 1h, 2h and 165h, and, (during target-controlled-infusion) 167h 35min, 167h 59min and 168h 25min after the burn injury
  The secondary hyperalgesia area is determined using a "weighted-pin" stimulator (PinPrick stimulators, MRC Systems GmbH, Heidelberg, Germany; 128 mN [2,606 kPa]). The borders of the areas are assessed by stimulating along eight symmetrical lines, converging towards the center of the burn injury. The stimulation path starts at least 12 cm outside the borders of the burn injury area. The participants are instructed to report, with their eyes closed, when the perception of the stimulus changes from an innocuous pin-prick to a stinging, smarting and unpleasant sensation, and the position is indicated by a marker.

SECONDARY OUTCOMES:
Pain during burn injury | Baseline, ½min, 1min, 2min, 3min, 4min, 5min, 6min and 7min during the burn injury
  Assessments are obtained by a visual analog rating scale (VAS)
Pin-prick pain thresholds (PPT) assessed by weighted-pin instruments at primary and secondary hyperalgesia areas | Baseline, 1h, 2h and 165h, and, (during target-controlled-infusion) 168h 25min after the burn injury
  Pin-prick pain thresholds (PPTs) in the primary BI-area and in the secondary hyperalgesia area are assessed by "weighted-pin" stimulators (8 to 512 mN [81 to 10,424 kPa]), starting with the lightest pin-prick stimulator (8 mN), and applying a modified Dixon's up-and-down technique. Participants are instructed to report the number of stimuli perceived as unpleasant after a total of five pin-prick stimuli. The lowest pinprick force associated with ≥ 3 unpleasant stimuli is defined as the PPT. The median value of the five PPTs is used in further data analysis. The PPT-data (8, 16, 32, 64, 128, 256, 512 mN) are converted to corresponding ordinal values 1 to 8, where the "cut-off" value of 8 is registered if no pain is elicited during assessment with the heaviest pin-prick stimulator (512 mN).
Online Reaction Time | Baseline, 1h, 2h and 165h, and, (during target-controlled-infusion) 167h 35min, 167h 59min and 168h 25min
  Online Reaction Time is measured using http://getyourwebsiteherecom/jswb/rttest01.htm. This computer-application shows a red-green traffic light. Participants are instructed to press the button when the light changes from red to green. Three measurements are used and the median value is used as a representative estimate of reaction time.
Clinical Opiate Withdrawal Scale (COWS) | Baseline and 165h, and, (during target-controlled-infusion) 167h 35min, 167h 59min and 168h 25min after the burn injury
  The Clinical Opiate Withdrawal Scale (COWS) is an examiner-based scale evaluating signs of opioid-withdrawal. Grading of symptoms, i.e. heart rate changes, sweating, restlessness, pupil size, bone or joint aches, running nose or tearing, nausea, vomiting, diarrhea, tremor, yawning, anxiety or irritability and "goose-flesh", are made in 11 categories. COWS-scores are divided into: 5-12 = mild; 13-24 = moderate; 25-36 = moderately severe ;> 36 = severe withdrawal reactions.
Hospital Anxiety and Depression Scale (HADS) | Baseline
  The Hospital Anxiety and Depression Scale (HADS) is used to assess anxiety and signs of depression. Based on 14 questions about the subject's status in the previous week, HADS measures agitation/anxiety and depression via two subscales (each containing seven questions). Participants have to answer each question on a scale of 0 to 3. The two subscales are summed separately. The maximum score of each subscale is 21 points and a score of 11 or more points suggests that the participant might be suffering from anxiety or depression. In case of score > 11 points in the depression subscale of the HADS, a physician will decide if there are clinical signs of depression. If there are signs of depression, this diagnosis will be told to the participant. The participant will be informed that the diagnosis of depression is based on clinical assessments - the HADS scale can be included in the diagnostic procedure. If it is the participants wish, he should visit his general practitioner for diagnosis
Pain Catastrophizing Scale (PCS) | Baseline
  The Pain Catastrophizing Scale (PCS) consists of 13 questions divided into three sections: rumination, exaggeration and helplessness. The questions are answered in accordance to a scale of 0 to 4. There is evidence of catastrophizing thoughts at a total score > 30 points.

CONTACTS AND LOCATIONS:
Overall Officials: Mads U Werner, MD, DMSc, Principal Investigator — Neuroscience Center, Copenhagen University Hospital, Denmark; Bradley K Taylor, M.Sc., Ph.D., Study Chair — Department of Physiology, University of Kentucky Medical Center
Locations (1):
- Neuroscience Center, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available

REFERENCES:
- [Background] Edwards RR, Ness TJ, Fillingim RB. Endogenous opioids, blood pressure, and diffuse noxious inhibitory controls: a preliminary study. Percept Mot Skills. 2004 Oct;99(2):679-87. doi: 10.2466/pms.99.2.679-687. PMID 15560360
- [Background] Taylor BK, Corder G. Endogenous analgesia, dependence, and latent pain sensitization. Curr Top Behav Neurosci. 2014;20:283-325. doi: 10.1007/7854_2014_351. PMID 25227929
- [Background] Werner MU, Pereira MP, Andersen LP, Dahl JB. Endogenous opioid antagonism in physiological experimental pain models: a systematic review. PLoS One. 2015 Jun 1;10(6):e0125887. doi: 10.1371/journal.pone.0125887. eCollection 2015. PMID 26029906
- [Result] Brennum J, Kaiser F, Dahl JB. Effect of naloxone on primary and secondary hyperalgesia induced by the human burn injury model. Acta Anaesthesiol Scand. 2001 Sep;45(8):954-60. doi: 10.1034/j.1399-6576.2001.450806.x. PMID 11576045
- [Result] Pielsticker A, Haag G, Zaudig M, Lautenbacher S. Impairment of pain inhibition in chronic tension-type headache. Pain. 2005 Nov;118(1-2):215-23. doi: 10.1016/j.pain.2005.08.019. Epub 2005 Oct 3. PMID 16202520
- [Result] Koppert W, Filitz J, Troster A, Ihmsen H, Angst M, Flor H, Schuttler J, Schmelz M. Activation of naloxone-sensitive and -insensitive inhibitory systems in a human pain model. J Pain. 2005 Nov;6(11):757-64. doi: 10.1016/j.jpain.2005.07.002. PMID 16275600
- [Result] Campillo A, Cabanero D, Romero A, Garcia-Nogales P, Puig MM. Delayed postoperative latent pain sensitization revealed by the systemic administration of opioid antagonists in mice. Eur J Pharmacol. 2011 Apr 25;657(1-3):89-96. doi: 10.1016/j.ejphar.2011.01.059. Epub 2011 Feb 4. PMID 21300053
- [Result] Corder G, Doolen S, Donahue RR, Winter MK, Jutras BL, He Y, Hu X, Wieskopf JS, Mogil JS, Storm DR, Wang ZJ, McCarson KE, Taylor BK. Constitutive mu-opioid receptor activity leads to long-term endogenous analgesia and dependence. Science. 2013 Sep 20;341(6152):1394-9. doi: 10.1126/science.1239403. PMID 24052307
- [Result] Pereira MP, Werner MU, Ringsted TK, Rowbotham MC, Taylor BK, Dahl JB. Does naloxone reinstate secondary hyperalgesia in humans after resolution of a burn injury? A placebo-controlled, double-blind, randomized, cross-over study. PLoS One. 2013 May 31;8(5):e64608. doi: 10.1371/journal.pone.0064608. Print 2013. PMID 23741350
- [Result] Pereira MP, Donahue RR, Dahl JB, Werner M, Taylor BK, Werner MU. Endogenous Opioid-Masked Latent Pain Sensitization: Studies from Mouse to Human. PLoS One. 2015 Aug 25;10(8):e0134441. doi: 10.1371/journal.pone.0134441. eCollection 2015. PMID 26305798
- [Result] Werner MU, Petersen KL, Rowbotham MC, Dahl JB. Healthy volunteers can be phenotyped using cutaneous sensitization pain models. PLoS One. 2013 May 9;8(5):e62733. doi: 10.1371/journal.pone.0062733. Print 2013. PMID 23671631